CLINICAL TRIAL: NCT02017028
Title: Correlation Between Endothelial Function and Trans Radial-procedural Events
Status: Withdrawn | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-13-0824-IB-CTIL
Record Dates: First submitted 2013-12-10; First posted 2013-12-20 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2016-05

CONDITIONS: Injury; Blood Vessel, Wrist, Radial Artery
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to investigate the relation between the previous presence of endothelial dysfunction and the development of radial artery vasospasm during the trans-radial coronary evaluation.

DETAILED DESCRIPTION:
All patient will undergo pre procedural endoPAT assessment for endothelial dysfunction

ELIGIBILITY:
Inclusion Criteria:

Patients without angiographic proof of coronary disease, with scheduled elective coronary angiographic evaluation by radial approach.

Exclusion Criteria:

Impossibility to perform radial approach; abnormal Barbeau test result (type C and D); previous important trauma of the upper limbs; presence of fistule for renal dialysis; lymphedema; acute myocardial infarction, severe valvular heart disease; patients with NYHA class III and IV heart failure; malignancy; active myocarditis; HIV infection or immunodeficiency state; chronic viral infection; acute systemic infection requiring antibiotics; systemic inflammatory disease; Raynaud's syndrome; refusal to sign the informed consent form. All participants must give a written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planned for elective trans-radial cath
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
To assess relation between the presence of previous endothelial dysfunction and radial artery vasospasm | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Amit Segev, MD, Principal Investigator — Sheba MC
Locations (1):
- Sheba Medical center, Ramat Gan, Israel